CLINICAL TRIAL: NCT04217044
Title: Histopathology Images Based Prediction of Molecular Pathology in Glioma Using Deep Learning or Machine Learning
Brief Title: Histopathology Images Based Prediction of Molecular Pathology in Glioma Using Artificial Intelligence
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhenyu Zhang, Principal Investigator, The First Affiliated Hospital of Zhengzhou University
Other Study IDs: GliomaAI-3
Record Dates: First submitted 2019-12-30; First posted 2020-01-03 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Glioma
Keywords: Molecular; Histopathology image; Deep Learning; Machine Learning
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 120 Months
Biospecimen Retention: Samples With DNA — All participants have signed the informed consent. Fresh frozen tissues of participants are collected immediately after tumor resection and preserved in liquid nitrogen. Whole exome sequencing, RNA sequencing and proteomics are planed to be conducted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Histopathology images based prediction of molecular pathology — Histopathology images based prediction of 1p/19q co-deletion, MGMT methylation, IDH and TERTp mutations or molecular subgroups by leveraging AI

SUMMARY:
This registry aims to collect clinical, molecular and radiologic data including detailed clinical parameters, molecular pathology (1p/19q co-deletion, MGMT methylation, IDH and TERTp mutations, etc) and images of HE slices in primary gliomas. By leveraging artificial intelligence, this registry will seek to construct and refine histopathology image based algorithms that are able to predict molecular pathology or subgroups of gliomas.

DETAILED DESCRIPTION:
Non-invasive and precise prediction for molecular biomarkers such as 1p/19q co-deletion, MGMT methylation, IDH and TERTp mutations is challenging. With the development of artificial intelligence, much more potential lies in the histopathology images of HE slices in primary gliomas could be excavated to aid prediction of molecular pathology of gliomas. The creation of a registry for primary glioma with detailed molecular pathology, histopathology image data and with sufficient sample size for deep learning (>1000) provide considerable opportunities for personalized prediction of molecular pathology with non-invasiveness and precision.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have radiologically and histologically confirmed diagnosis of primary glioma
* Life expectancy of greater than 3 months
* Must receive tumor resection
* Signed informed consent

Exclusion Criteria:

* No gliomas
* No sufficient amount of tumor tissues for detection of molecular pathology
* Patients who are pregnant or breast feeding
* Patients who are suffered from severe systematic malfunctions

Ages: 1 Year to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with newly diagnosed glioma that receive tumor resection
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
AUC of prediction performance | up to 10 years
  AUC=sensitivity+specificity-1

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided
Undecided